CLINICAL TRIAL: NCT05904249
Title: Investigation of the Effectiveness of Telerehabilitation in Individuals With Rotator Cuff Tear
Brief Title: Telerehabilitation in Individuals With Rotator Cuff Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Emrah Zirek, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IstanbulU
Record Dates: First submitted 2022-03-02; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Rotator Cuff Tears; Physiotherapy and Rehabilitation; Shoulder Pain; Rotator Cuff Injuries
Keywords: Telerehabilitation; Remote Rehabilitations; Exercise Therapy; Telemedicine
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study groups will be randomized by Researcher 3 using the Research Randomizer (https://www.randomizer.org). Researcher 1 will be blinded when selecting a treatment group.
  Rehabilitation practices for both groups will be conducted by the Researcher 1 and outcome evaluation will be conducted by the Researcher 2. The Researcher 2 will not know which group the data of the patient he/she is evaluating belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet Based Synchronized Telerehabilitation Group (Group 1) (Experimental): The treatments of the participants who meet the inclusion criteria in the study will be conducted remotely via instant video communication. The Specialist Physiotherapist will apply the necessary exercises, verbal guidance or repetition of the movements shown, according to the patient's condition, synchronized via instant video and audio calls (Whatsapp or Zoom).
  Interventions: Other: Internet Based Synchronized Telerehabilitation
- Face-to-Face Rehabilitation Group (Group 2) (Experimental): The treatments of the participants that meet the inclusion criteria of the study will be administered by Specialist Physiotherapist. The progress of the patients will be regularly followed up on a weekly basis, and treatments will be applied in accordance with the program in rehabilitation.
  Interventions: Other: Face-to-Face Rehabilitation

INTERVENTIONS:
Other: Internet Based Synchronized Telerehabilitation — Week 1
  * Posterior capsule stretching
  * Passive range of motion
  * Wand exercises in supine position
  * Scapular adduction exercise
  * Ball rolling on the table (<90°)
  * Coldpack (15min)
  Week 2
  * Wand exercises while standing.
  * Ball roll on wall (>90°)
  * Ball roll on the table (90°)
  * Weightless External Rotation exercises
  * Functional PNF movements
  Week 3
  * Resistive scapulothoracic strengthening
  * Ball scrolling on the table (resistive)
  Week 4
  * Single handed ball roll on the table (>90°)
  * External rotation exercise with 0.5-1kg weight in side lying
  * Strengthening exercises, shoulder in 90° scapulation for 10s
  Week 5
  * External rotation with 0.5-1 kg weight in side lying
  * Strengthening exercises by keeping the shoulder in 90° scapulation for 10s
  Week 6-8
  * Dynamic hugs and push up plus
  * Ball throwing and catching
  Arms: Internet Based Synchronized Telerehabilitation Group (Group 1)
Other: Face-to-Face Rehabilitation — Week 1
  * Posterior capsule stretching
  * Passive range of motion
  * Wand exercises in supine position
  * Scapular adduction exercise
  * Ball rolling on the table (<90°)
  * Coldpack (15min)
  Week 2
  * Wand exercises while standing.
  * Ball roll on wall (>90°)
  * Ball roll on the table (90°)
  * Weightless External Rotation exercises
  * Functional PNF movements
  Week 3
  * Resistive scapulothoracic strengthening
  * Ball scrolling on the table (resistive)
  Week 4
  * Single handed ball roll on the table (>90°)
  * External rotation exercise with 0.5-1kg weight in side lying
  * Strengthening exercises, shoulder in 90° scapulation for 10s
  Week 5
  * External rotation with 0.5-1 kg weight in side lying
  * Strengthening exercises by keeping the shoulder in 90° scapulation for 10s
  Week 6-8
  * Dynamic hugs and push up plus
  * Ball throwing and catching
  Arms: Face-to-Face Rehabilitation Group (Group 2)

SUMMARY:
The majority of patients presenting with shoulder pain are those with rotator cuff problems. Although telerehabilitation is a promising field in many areas, there is still limited high-quality research with strong evidence of its effectiveness for musculoskeletal problems. In this study, online rehabilitation and face-to-face rehabilitation will be compared in people with partial rotator cuff tears.

DETAILED DESCRIPTION:
The prevalence of shoulder pain increases with age and is mostly associated with inadequate treatment of symptoms. A large part of the patients who apply to the clinic with the complaint of shoulder pain are individuals with rotator cuff problems. Partial rotator cuff (RM) tear is defined as tears that can be seen on the superior, inferior, or both sides of the cuff. It is stated that the most critical risk factors for RM tear are age, dominant arm, and trauma. The degenerative process is generally considered normal in age-related tears and is seen in 20% of individuals over the age of 65.

The Coronavirus disease (COVID-19), is still the most important global concern. People with chronic diseases have been known to delay getting healthcare services due to fear of the risk of infection following the COVID-19 pandemic. This could lead to increased morbidity and mortality due to delay and disruption in access to treatment applications needed for patient populations other than COVID-19. At this stage, one of the applications that can be effective for disturbed patient healing processes is the Telerehabilitation application, which has proven its effectiveness in previous epidemics (EBOLA, SARS, etc.), when patients are treated remotely after and after treatment. Especially during the COVID-19 pandemic, there has been an increase in the need for Internet-based remote treatment approaches, as it allows both patients and physiotherapists to advance the treatment process without the risk of infection. In the next decade, telerehabilitation options are expected to diversify and become widespread in assessing and treating many diseases with emerging technologies.

Studies have shown that despite the growing number of applications of telerehabilitation worldwide, evidence for clinical effectiveness is still limited. In addition, the effectiveness of telerehabilitation for musculoskeletal problems has not been fully demonstrated due to the lack of a specific standard for telerehabilitation and the variability of the approaches used. In conclusion, although telerehabilitation is a promising field in many areas, there is still a limited amount of good-quality research with strong evidence.

Therefore, this study aimed to compare the effects of internet-based telerehabilitation and face-to-face rehabilitation practices on pain, range of motion, functionality, and quality of life in patients with partial rotator cuff injury.

ELIGIBILITY:
Inclusion Criteria:

* Presence of bursal facial tear 1 cm below the tear degree; presence of complaints of shoulder pain lasting for a minimum of 1 and a maximum of 6 months; having been diagnosed with partial rotator cuff tear by an orthopedist who is an expert in the field; no shoulder instability; inadequate response to non-operative treatment (corticosteroid injection, anti-inflammatory drugs, rest and physiotherapy and rehabilitation); not using corticosteroid drug; being between the ages of 18-60; to have sufficient knowledge, skills and technological tools to access the Tele-Rehabilitation application.

Exclusion Criteria:

* Presence of malignancy affecting the shoulder region; disc herniations that may cause shoulder pain; individuals with inflammatory joint disease; osteoarthritis of the humeral head; history of surgery affecting the shoulder; inability of the patient to cooperate; systemic problems that cannot be controlled with medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | One year
  Patients' pain levels at rest, during activity, and at night will be assessed using a Visual Analog Scale (VAS). The score is determined by measuring the distance (mm) on a 10 cm line between the "no pain" anchor and the patient's mark, providing a score range of 0 to 100. A higher score indicates greater pain intensity.
Range of Motion Assessment | One year
  The range of motion values of the participants will be recorded using the universal goniometer, which is an objective tool used in clinical range of motion measurement.The flexion, scapular abduction, internal and external rotation values of the shoulder joint will be measured in the supine position with a universal goniometer in accordance with the procedure in the literature.
Muscle Activation Assessment | One year
  Delsys Biometrics Datalite WS450, a surface EMG system, will be used to evaluate the function of the shoulder muscles. Previous studies and the website of the SENIAM project of the European Union Biomedical Health and Research Program (http://www.seniam.org/) will be accepted as reference.
The Disabilities of the Arm, Shoulder and Hand Questionnaire | One year
  Hand, Shoulder and Hand Disability Questionaire will be used to assess the functional state of the participants. The possible score ranges from 0 to 100 points. 0 points represent full unrestricted upper limb function and 100 points represent the maximum possible functional impairment.
American Standardized Shoulder and Elbow Surgeon Assessment Form | One year
  The ASES section on patient self-reports is a condition-specific scale, i.e. it is for a specific condition that is intended to measure functional limitation and shoulder pain. The total pain score and the functional score are equally weighted (50 points each) and are combined to obtain a total score out of a possible 100 points.
Modified Constant-Murley | One year
  The Modified Constant-Murley Scale is widely used to assess disability associated with shoulder injuries, but has been criticized for its use of inaccurate terminology and the lack of a standardized methodology. The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. The higher the score, the higher the quality of the function.

SECONDARY OUTCOMES:
Short Form-12 | One year
  Short Form-12 will be used to assess quality of life related to physical and mental health. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). SF-12 PCS mean scores ranged between 48.3 and 49.2, and SF-12 MCS mean scores ranged between 48.0 and 49.6.
Global Change Scale | One year
  The satisfaction levels of the participants will be assessed using the Global Change Scale. Subjects are asked to rate their post-treatment status on a 5-point scale (-2: I am much worse, -1: I am worse, 0: I am the same, 1: I am better, 2: I am much better). A high score is considered a sign of high satisfaction.
Hospital Anxiety and Depression Scale | One year
  Participants' levels of anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale. The Hospital Anxiety and Depression Scale is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21); 0-7 (Normal) 8-10 (Mild) 11-15 (Moderate) 16-21 (Severe).

CONTACTS AND LOCATIONS:
Overall Officials: Nuri Aydin, Prof.Dr, Study Chair — Istanbul University - Cerrahpasa; Mehmet Fatih Guven, Assoc.Prof., Study Chair — Istanbul University - Cerrahpasa; Emrah Zirek, Res.Assist., Principal Investigator — Bingol University; Yildiz Analay Akbaba, Assoc.Prof., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpasa, Faculty of Medicine, Department of Orthopedics and Traumatology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agostini M, Moja L, Banzi R, Pistotti V, Tonin P, Venneri A, Turolla A. Telerehabilitation and recovery of motor function: a systematic review and meta-analysis. J Telemed Telecare. 2015 Jun;21(4):202-13. doi: 10.1177/1357633X15572201. Epub 2015 Feb 22. PMID 25712109
- [Background] Ainsworth R, Lewis JS. Exercise therapy for the conservative management of full thickness tears of the rotator cuff: a systematic review. Br J Sports Med. 2007 Apr;41(4):200-10. doi: 10.1136/bjsm.2006.032524. Epub 2007 Jan 30. PMID 17264144
- [Background] Assad-Uz-Zaman, M., Islam, M. R., Rahman, M. H., Wang, Y. C., & McGonigle, E.. Kinect controlled NAO robot for telerehabilitation. Journal of Intelligent Systems, 20213; 0(1), 224-239.
- [Background] Berton A, Longo UG, Candela V, Fioravanti S, Giannone L, Arcangeli V, Alciati V, Berton C, Facchinetti G, Marchetti A, Schena E, De Marinis MG, Denaro V. Virtual Reality, Augmented Reality, Gamification, and Telerehabilitation: Psychological Impact on Orthopedic Patients' Rehabilitation. J Clin Med. 2020 Aug 7;9(8):2567. doi: 10.3390/jcm9082567. PMID 32784745
- [Background] Boykin, R. E., Heuer, H. J., Vaishnav, S., & Millett, P. J. Rotator cuff disease-basics of diagnosis and treatment. Rheumatology Reports, 2010; 2(1), e1-e1.
- [Background] Carlsson AM. Assessment of chronic pain. I. Aspects of the reliability and validity of the visual analogue scale. Pain. 1983 May;16(1):87-101. doi: 10.1016/0304-3959(83)90088-X. PMID 6602967
- [Background] Contreras CM, Metzger GA, Beane JD, Dedhia PH, Ejaz A, Pawlik TM. Telemedicine: Patient-Provider Clinical Engagement During the COVID-19 Pandemic and Beyond. J Gastrointest Surg. 2020 Jul;24(7):1692-1697. doi: 10.1007/s11605-020-04623-5. Epub 2020 May 8. PMID 32385614
- [Background] Celik D. Turkish version of the modified Constant-Murley score and standardized test protocol: reliability and validity. Acta Orthop Traumatol Turc. 2016;50(1):69-75. doi: 10.3944/AOTT.2016.14.0354. PMID 26854052
- [Background] Celik D, Atalar AC, Demirhan M, Dirican A. Translation, cultural adaptation, validity and reliability of the Turkish ASES questionnaire. Knee Surg Sports Traumatol Arthrosc. 2013 Sep;21(9):2184-9. doi: 10.1007/s00167-012-2183-3. Epub 2012 Aug 30. PMID 22932692
- [Background] Danhieux K, Buffel V, Pairon A, Benkheil A, Remmen R, Wouters E, van Olmen J. The impact of COVID-19 on chronic care according to providers: a qualitative study among primary care practices in Belgium. BMC Fam Pract. 2020 Dec 5;21(1):255. doi: 10.1186/s12875-020-01326-3. PMID 33278877
- [Background] Diercks R, Bron C, Dorrestijn O, Meskers C, Naber R, de Ruiter T, Willems J, Winters J, van der Woude HJ; Dutch Orthopaedic Association. Guideline for diagnosis and treatment of subacromial pain syndrome: a multidisciplinary review by the Dutch Orthopaedic Association. Acta Orthop. 2014 Jun;85(3):314-22. doi: 10.3109/17453674.2014.920991. Epub 2014 May 21. PMID 24847788
- [Background] Dominguez-Romero JG, Jimenez-Rejano JJ, Ridao-Fernandez C, Chamorro-Moriana G. Exercise-Based Muscle Development Programmes and Their Effectiveness in the Functional Recovery of Rotator Cuff Tendinopathy: A Systematic Review. Diagnostics (Basel). 2021 Mar 16;11(3):529. doi: 10.3390/diagnostics11030529. PMID 33809604
- [Background] Düger, T., Yakut, E., Öksüz, Ç., Yörükan, S., Bilgütay, B. S., Ayhan, Ç., . . . Yakut, Y. (2006). Kol, omuz ve el sorunları (disabilities of the arm, shoulder and hand-DASH) anketi Türkçe uyarlamasının güvenirliği ve geçerliği. Fizyoterapi Rehabilitasyon, 17(3), 99-107.
- [Background] Edwards P, Ebert J, Joss B, Bhabra G, Ackland T, Wang A. EXERCISE REHABILITATION IN THE NON-OPERATIVE MANAGEMENT OF ROTATOR CUFF TEARS: A REVIEW OF THE LITERATURE. Int J Sports Phys Ther. 2016 Apr;11(2):279-301. PMID 27104061
- [Background] Edwards PK, Ebert JR, Littlewood C, Ackland T, Wang A. A Systematic Review of Electromyography Studies in Normal Shoulders to Inform Postoperative Rehabilitation Following Rotator Cuff Repair. J Orthop Sports Phys Ther. 2017 Dec;47(12):931-944. doi: 10.2519/jospt.2017.7271. Epub 2017 Jul 13. PMID 28704624
- [Background] Erdfelder, E., Faul, F., & Buchner, A. GPOWER: A general power analysis program. Behavior Research Methods, Instruments, & Computers, 1996; 28(1), 1-11. doi:10.3758/BF03203630
- [Background] Franchignoni F, Vercelli S, Giordano A, Sartorio F, Bravini E, Ferriero G. Minimal clinically important difference of the disabilities of the arm, shoulder and hand outcome measure (DASH) and its shortened version (QuickDASH). J Orthop Sports Phys Ther. 2014 Jan;44(1):30-9. doi: 10.2519/jospt.2014.4893. Epub 2013 Oct 30. PMID 24175606
- [Background] Gava V, Ribeiro LP, Barreto RPG, Camargo PR. Effectiveness of physical therapy given by telerehabilitation on pain and disability of individuals with shoulder pain: A systematic review. Clin Rehabil. 2022 Jun;36(6):715-725. doi: 10.1177/02692155221083496. Epub 2022 Mar 1. PMID 35230167
- [Background] Hailey D, Roine R, Ohinmaa A, Dennett L. Evidence of benefit from telerehabilitation in routine care: a systematic review. J Telemed Telecare. 2011;17(6):281-7. doi: 10.1258/jtt.2011.101208. Epub 2011 Aug 15. PMID 21844172
- [Background] Hill CL, Gill TK, Shanahan EM, Taylor AW. Prevalence and correlates of shoulder pain and stiffness in a population-based study: the North West Adelaide Health Study. Int J Rheum Dis. 2010 Aug;13(3):215-22. doi: 10.1111/j.1756-185X.2010.01475.x. PMID 20704617
- [Background] Holmgren T, Hallgren HB, Oberg B, Adolfsson L, Johansson K. Effect of specific exercise strategy on need for surgery in patients with subacromial impingement syndrome: randomised controlled study. Br J Sports Med. 2014 Oct;48(19):1456-7. doi: 10.1136/bjsports-2014-e787rep. PMID 25213604
- [Background] Itoi E, Tabata S. Conservative treatment of rotator cuff tears. Clin Orthop Relat Res. 1992 Feb;(275):165-73. PMID 1735208
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Katz, N. B., & Tenforde, A. S. Telerehabilitation for Musculoskeletal Injuries. In Telerehabilitation 2022; (pp. 197-212). Elsevier.
- [Background] Koçyiğit, H., Aydemir, Ö., Fişek, G., Ölmez, N., & Memiş, A. K. Form-36 (KF-36)'nın Türkçe versiyonunun güvenilirliği ve geçerliliği. Ilaç ve tedavi dergisi, 1999; 12(2), 102-106.
- [Background] Michener LA, McClure PW, Karduna AR. Anatomical and biomechanical mechanisms of subacromial impingement syndrome. Clin Biomech (Bristol). 2003 Jun;18(5):369-79. doi: 10.1016/s0268-0033(03)00047-0. PMID 12763431
- [Background] Ohannessian R, Duong TA, Odone A. Global Telemedicine Implementation and Integration Within Health Systems to Fight the COVID-19 Pandemic: A Call to Action. JMIR Public Health Surveill. 2020 Apr 2;6(2):e18810. doi: 10.2196/18810. PMID 32238336
- [Background] Otman, A. S. Tedavi hareketlerinde temel değerlendirme prensipleri Pelikan yayıncılık. 2014; pp: 66-70
- [Background] Pallant, J. SPSS survival manual: A step by step guide to data analysis using IBM SPSS. Routledge.2020
- [Background] Pastora-Bernal JM, Martin-Valero R, Baron-Lopez FJ. Cost analysis of telerehabilitation after arthroscopic subacromial decompression. J Telemed Telecare. 2018 Sep;24(8):553-559. doi: 10.1177/1357633X17723367. Epub 2017 Aug 17. PMID 28816578
- [Background] Pastora-Bernal JM, Martin-Valero R, Baron-Lopez FJ, Estebanez-Perez MJ. Evidence of Benefit of Telerehabitation After Orthopedic Surgery: A Systematic Review. J Med Internet Res. 2017 Apr 28;19(4):e142. doi: 10.2196/jmir.6836. PMID 28455277
- [Background] Powell JK, Schram B, Lewis J, Hing W. Physiotherapists nearly always prescribe exercise for rotator cuff-related shoulder pain; but why? A cross-sectional international survey of physiotherapists. Musculoskeletal Care. 2023 Mar;21(1):253-263. doi: 10.1002/msc.1699. Epub 2022 Sep 11. PMID 36089802
- [Background] Rogante M, Grigioni M, Cordella D, Giacomozzi C. Ten years of telerehabilitation: A literature overview of technologies and clinical applications. NeuroRehabilitation. 2010;27(4):287-304. doi: 10.3233/NRE-2010-0612. PMID 21160118
- [Background] Sgroi TA, Cilenti M. Rotator cuff repair: post-operative rehabilitation concepts. Curr Rev Musculoskelet Med. 2018 Mar;11(1):86-91. doi: 10.1007/s12178-018-9462-7. PMID 29399735
- [Background] Stawicki SP, Jeanmonod R, Miller AC, Paladino L, Gaieski DF, Yaffee AQ, De Wulf A, Grover J, Papadimos TJ, Bloem C, Galwankar SC, Chauhan V, Firstenberg MS, Di Somma S, Jeanmonod D, Garg SM, Tucci V, Anderson HL, Fatimah L, Worlton TJ, Dubhashi SP, Glaze KS, Sinha S, Opara IN, Yellapu V, Kelkar D, El-Menyar A, Krishnan V, Venkataramanaiah S, Leyfman Y, Saoud Al Thani HA, Wb Nanayakkara P, Nanda S, Cioe-Pena E, Sardesai I, Chandra S, Munasinghe A, Dutta V, Dal Ponte ST, Izurieta R, Asensio JA, Garg M. The 2019-2020 Novel Coronavirus (Severe Acute Respiratory Syndrome Coronavirus 2) Pandemic: A Joint American College of Academic International Medicine-World Academic Council of Emergency Medicine Multidisciplinary COVID-19 Working Group Consensus Paper. J Glob Infect Dis. 2020 May 22;12(2):47-93. doi: 10.4103/jgid.jgid_86_20. eCollection 2020 Apr-Jun. PMID 32773996
- [Background] Turolla A, Rossettini G, Viceconti A, Palese A, Geri T. Musculoskeletal Physical Therapy During the COVID-19 Pandemic: Is Telerehabilitation the Answer? Phys Ther. 2020 Aug 12;100(8):1260-1264. doi: 10.1093/ptj/pzaa093. No abstract available. PMID 32386218
- [Background] Turkmen E, Analay Akbaba Y, Altun S. Effectiveness of video-based rehabilitation program on pain, functionality, and quality of life in the treatment of rotator cuff tears: A randomized controlled trial. J Hand Ther. 2020 Jul-Sep;33(3):288-295. doi: 10.1016/j.jht.2019.08.004. Epub 2020 Mar 17. PMID 32197805
- [Background] Wang S, Chapple CM, Quinn D, Tumilty S, Ribeiro DC. Dosage of joint mobilisation for the management of rotator cuff-related shoulder pain: protocol for a scoping review. BMJ Open. 2022 Jun 3;12(6):e056771. doi: 10.1136/bmjopen-2021-056771. PMID 36691247
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Xie Y, Szeto GP, Dai J, Madeleine P. A comparison of muscle activity in using touchscreen smartphone among young people with and without chronic neck-shoulder pain. Ergonomics. 2016;59(1):61-72. doi: 10.1080/00140139.2015.1056237. Epub 2015 Jul 28. PMID 26218600
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Derived] Zirek E, Analay Akbaba Y, Guven MF. Is synchronous telerehabilitation effective in the treatment of rotator cuff tears? - a randomized controlled trial. Physiother Theory Pract. 2025 Dec;41(12):2501-2512. doi: 10.1080/09593985.2025.2526021. Epub 2025 Jul 2. PMID 40601531